CLINICAL TRIAL: NCT02191397
Title: A Multi-centre, Randomised, Double-blind, Parallel Active-controlled Study Evaluating the Efficacy, Safety and Tolerability of Bupropion Hydrochloride Extended-release (Bupropion XL 300mg Once Daily), Escitalopram Oxalate (Escitalopram, 10mg-20mg Once Daily) in Subjects With Major Depressive Disorder
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of Bupropion Hydrochloride Extended-release Tablet, and Escitalopram Oxalate Capsule in Subjects With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114589
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder, Major
Keywords: Escitalopram; Major depressive disorder; Non-inferiority; Bupropion
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupropion Treatment Arm (Experimental): Subject will receive bupropion in 3 dose levels along with escitalopram matching placebo to maintain the blind in acute treatment phase. At dose level 1 (Week 0 to Week 1), Subjects will receive bupropion XL 150 milligram (mg) per day for a week. At dose level 2 (Week 1 to Week 4), bupropion XL dose will be increased to 300mg/day for further 3 weeks. At dose level 3 (Week 4 to Week 8), bupropion XL dose will be maintained at 300mg/day. Subjects intolerable to dose level 3 will be allowed to down titrate to dose level 2 at anytime, and maintain the dose until the end of acute treatment phase (Week 8, Visit 7). At the end of acute treatment phase, the dose of bupropion XL will be reduced to 150mg/day for 1 week before discontinuation.
  Interventions: Drug: Bupropion; Drug: Escitalopram Matching Placebo
- Escitalopram Treatment Arm (Active Comparator): Subject will receive escitalopram in 3 dose levels along with bupropion matching placebo to maintain the blind in acute treatment phase. At dose level 1 (Week 0 to Week 1), Subjects will receive escitalopram 10mg/day for a week. At dose level 2 (Week 1 to Week 4), escitalopram dose will be maintained at 10mg/day for further 3 weeks. At dose level 3 (Week 4 to Week 8), escitalopram dose will be increased to 20mg/day. Subjects intolerable to dose level 3 will be allowed to down titrate to dose level 2 at anytime, and maintain the dose until the end of acute treatment phase (Week 8, Visit 7). At the end of acute treatment phase, the dose of escitalopram 20mg/day, the dose will be reduced to 10 mg/day for 1 week before discontinuation, while those receiving 10mg/day will discontinuation directly.
  Interventions: Drug: Bupropion Matching Placebo; Drug: Escitalopram

INTERVENTIONS:
Drug: Bupropion — Bupropion is an extended-release plain creamy white colored tablet which contains bupropion hydrochloride equivalent to 150 mg of bupropion.
  Arms: Bupropion Treatment Arm
Drug: Bupropion Matching Placebo — Bupropion hydrochloride matching placebo tablets will be supplied to maintain blinding
  Arms: Escitalopram Treatment Arm
Drug: Escitalopram — Escitalopram is available as a Swedish orange capsule containing escitalopram oxalate equivalent to 10 mg of escitalopram.
  Arms: Escitalopram Treatment Arm
Drug: Escitalopram Matching Placebo — Escitalopram oxalate matching placebo tablets will be supplied to maintain blinding
  Arms: Bupropion Treatment Arm

SUMMARY:
This multi-centre study will follow a randomised, double-blind, parallel-group, active-controlled design and will evaluate the efficacy, safety and tolerability of bupropion extended-release (XL) (300 mg/day) compared with escitalopram (10-20 mg/day) in outpatients and inpatients with major depressive disorder (MDD). The total duration of the study will be 11 weeks consisting of three phases. The screening phase (phase I) will be lasting for 0-14 days, subjects will be randomised to bupropion XL or escitalopram in a 1:1 ratio for acute phase treatment phase (phase II) for 8 weeks. There are 3 dose levels during this acute treatment phase. The 3-dose level plan is designed to ensure each drug is titrated according to the prescribing information and to reach an optimal clinical dose. Finally patients will enter the taper phase (phase III) for up to 1 week to assess and reduce the possible withdrawal symptoms.

In China almost all existing antidepressants are available on the market, but bupropion XL has not yet been approved. This Phase III clinical trial will be used for the purpose of registering bupropion XL in China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to effectively communicate with investigator, complete study related documents, comprehend the key components of the consent form and must provide written informed consent to participate in the study prior to any study-specific assessments or procedures.
* An in- patient or out-patient (male or female) and aged >=18 years.
* A diagnosis of MDD, nonpsychotic, single episode or recurrent, Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) (296.2/296.3), utilizing the Mini International Neuropsychiatric Interview (MINI).
* Established MDD diagnosis with a duration of at least 4 weeks.
* HAMD-17 total score of >=20 and a CGI-S score of >=4 at both the Screening Visit and the Baseline Visit.
* Subject must be in general good health and be considered clinically appropriate for therapy with bupropion or escitalopram, based upon the investigator's overall clinical evaluation.
* Female patients of child-bearing potential only: patients must not be lactating and must test negative for pregnancy at screening and agree to use a medically accepted method of birth control during the study.
* Liver function tests: alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT (QTc) criteria： QTc <450 milliseconds (msec) or QTc <480msec for patients with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or machine or manual overread. For subject eligibility and withdrawal, QTcF will be used. For purpose of data analysis, QTcF will be used. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.

Exclusion Criteria:

* Has been diagnosed or received treatment for a primary Axis I disorder with the exception of MDD (including current or past diagnosis of anorexia nervosa or bulimia). Additionally, subjects diagnosed with dysthymic disorder within the past 2 years will be excluded.
* Current DSM-IV Axis II diagnosis that suggests non-compliance with the protocol.
* A subject who, in the assessment with the Columbia Suicide Severity Rating Scale (C-SSRS) and investigator's judgment, poses suicidal risk, or had suicide attempt or behavior within 6 months prior to the Screening Visit.
* Current or past history of seizure disorder or brain injury (traumatic or disease related); or any condition which, in the opinion of the investigator, predisposed to seizure; subjects treated with other medications or treatment regimes that lower seizure threshold. Note: single childhood febrile seizure is not exclusionary.
* In the Investigator's judgment, presence of clinically significant laboratory test results (including ECG, hematology, chemistry and urine), or the conditions which render patients unsuitable for the study (such as serious cardiovascular disease, uncontrolled hypertension, liver or renal insufficiency) and pose a safety concern or interfere with the accurate safety and efficacy assessments. Subjects with co-morbidities (such as diabetes, hypertension, hypothyroid, chronic respiratory diseases or other physical illness) were eligible if their condition had been stable for at least three months and they had been receiving standard therapy for the condition for at least three months.
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Frequent and/or severe allergic reactions with multiple medications, or history of a medically significant adverse effect (including allergic reaction) from any medications or compounds in the study.
* Use of prohibited psychotropic drugs not allowed within seven days (14 days for monoamine oxidase inhibitors (MAOIs), 30 days for fluoxetine) prior to the Baseline Visit.
* Subjects who have attended any studies investigating bupropion or escitalopram 6 months prior to this study, or use of bupropion or escitalopram in the last 4 weeks.
* Participation in other clinical studies unrelated to the current illness within 30 days or participation in other clinical studies related to the current illness within 3 months.
* Initiation of systematic psychotherapy within three months prior to the Screening Visit, or plans to initiate systematic psychotherapy during the study.
* Received electroconvulsive therapy (ECT), modify electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), or other physical therapy within the 6 months prior to the Screening Visit.
* Previous failure of bupropion or escitalopram treatment with adequate courses and doses.
* Previous or present failure of two different classes of antidepressants treatment with adequate courses (e.g. maximum labelled doses for >=4 weeks).
* History of substance abuse (alcohol or drugs) or substance dependence within 12 months (as defined in the DSM-IV).
* Other conditions which, in the Investigator's judgment, render patients unsuitable for the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- China (17):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Guiyang, Guizhou
  - GSK Investigational Site, Baoding, Hebei
  - GSK Investigational Site, Harbin, Heilongjiang
  - GSK Investigational Site, Changshacun, Henan
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Xi’an, Shanxi
  - GSK Investigational Site, Kunming, Yunnan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20102

REFERENCES:
- [Background] Shen Y, Zhao Q, Yu Y, Tan Y, Zhang H, Xu X, Wang Z, Li Y, Hu J, Zhong J, Li H. Efficacy and safety of bupropion hydrochloride extended-release versus escitalopram oxalate in Chinese patients with major depressive disorder: Results from a randomized, double-blind, non-inferiority trial. J Affect Disord. 2019 Oct 1;257:143-149. doi: 10.1016/j.jad.2019.07.023. Epub 2019 Jul 5. PMID 31301615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, randomized, double-blind, parallel active-controlled study to evaluate the efficacy, safety and tolerability of bupropion hydrochloride extended-release (XL) and escitalopram oxalate in participants with major depressive disorder. This study was conducted in China from 10-February-2015 to 25-October-2016.
Pre-assignment Details: The study had screening phase (up to 14 days), 8-week double blind treatment phase and taper phase (up to 1 week). A total of 655 participants were screened and 538 were randomized into the study. 4 participants were randomized but discontinued prior to receiving any study treatment. Hence, the Safety Population was comprised of 534 participants.
Groups:
- Bupropion XL: In a double-blind 8-week acute treatment phase, participants received 1 tablet of bupropion XL 150 milligram (mg) per day at dose level 1 (Week 0 to Week 1). At dose level 2 (Week 1 to Week 4), bupropion XL dose was increased to 300 mg per day (2 tablets of bupropion XL 150 mg) for further 3 weeks to ensure that participants had achieved the clinical recommended dose. At dose level 3 (Week 4 to Week 8), bupropion XL dose was still maintained at 300 mg per day (2 tablets of bupropion XL 150 mg). To ensure study blind, the participants were dosed with placebo matching escitalopram at each dose level. After treatment phase, participants entered in taper phase where dose in was down-titrated step by step to reduce the possible withdrawal symptoms. In taper phase, both dose level 2 and dose level 3 were down titrated to dose level 1 for 1 week before discontinuation.
- Escitalopram: In a double-blind 8-week acute treatment phase, participants received 1 capsule of escitalopram 10 mg per day at dose level 1 (Week 0 to Week 1). Escitalopram dose was maintained at 10 mg per day (1 capsule of Escitalopram 10 mg) for further 3 weeks to ensure that participants had achieved the clinical recommended dose. At dose level 3 (Week 4 to Week 8), the escitalopram dose could be increased to 20 mg per day (2 capsule of Escitalopram 10 mg). To ensure study blind, the participants were also dosed with placebo matching bupropion XL at each dose level. After treatment phase, participants entered in taper phase where dose in was down-titrated step by step to reduce the possible withdrawal symptoms. In taper phase, both dose level 2 and dose level 3 were down titrated to dose level 1 for 1 week before discontinuation.
Period: Overall Study
Arm/Group | Bupropion XL | Escitalopram
Started | 266 | 268
Completed | 183 | 198
Not Completed | 83 | 70
Not completed — Adverse Event | 28 | 17
Not completed — Lack of Efficacy | 10 | 5
Not completed — Protocol Violation | 0 | 3
Not completed — Met protocol-defined stopping criteria | 5 | 4
Not completed — Lost to Follow-up | 10 | 11
Not completed — Physician Decision | 8 | 3
Not completed — Withdrawal by Subject | 22 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion XL | Escitalopram | Total
Number analyzed (Participants) | 266 | 268 | 534
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (11.92) | 37.6 (12.09) | 37.3 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 172 | 340
  Male | 98 | 96 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 266 | 268 | 534

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hamilton Depression Rating Scale - 17 (HAMD-17) Total Score From Baseline to End of Acute Treatment Phase (Week 8)
Description: HAMD-17 is used to assess the severity of depression and symptom improvement. It consisted of 17 questions. The HAMD-17 total score is calculated by summing the individual response scores if there is no missing response. HAMD-17 has a total score in a range of 0 (not present) to 52 (severe). Change from Baseline was calculated by subtracting the Baseline total score (at Day 0, Week 0) from Week 8 observed total score. The Per Protocol (PP) Population is defined as all randomized participants in the Intent-To-Treat (ITT) Population who do not meet criteria of a major protocol deviation, with overall compliance of active drug for acute treatment phase in the range of 75%-125% and complete the first 6 weeks treatment and has HAMD-17 assessment at/after week 6 (that is >=35 days). All participants in the PP population were included in the mixed model repeated measures analysis. Only those participants with data available at the specified time point were analyzed.
Time Frame: Baseline (Week 0) and Week 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 176 | 188
Scores on a scale | -14.5 (0.41) | -15.4 (0.39)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Non-Inferiority — A one-sided 97.5% confidence interval for the between-treatment difference (bupropion XL-escitalopram) was compared with the pre-defined non-inferiority margin of 2.2. If the upper limit of the one-sided 97.5% confidence interval was below 2.2, then it indicated that bupropion was not inferior in efficacy to escitalopram; p = 0.139, Mixed model repeated measures analysis — Analysis included Baseline HAMD-17 total score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.27 to 1.94] — Observed Cases (OC) dataset was used, where available data at a given time point was used with no missing values filled in with estimates

2. Secondary Outcome: Response Rate Based on HAMD-17 Total Score
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 total score is calculated by summing the individual response scores if there is no missing response. HAMD-17 has a total score in a range of 0 (not present) to 52 (severe). Values at Day 0, Week 0 was considered as Baseline value. Response was defined as decrease in HAMD-17 total scores at end of acute treatment phase (Week 8) relative to Baseline by at least 50%. Non-responder Imputation was used in calculation of rates.
Time Frame: Up to Week 8
Population: PP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Percentage of Participants | 69.6 | 72.9
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.479, GEE model — P-value was estimated from a Generalized Estimating Equation (GEE) model with Response based on HADM-17 as response variable and treatment, gender as explanatory variables; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.55 to 1.33]

3. Secondary Outcome: Remission Rate Based on HAMD-17 Total Score
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 total score is calculated by summing the individual response scores if there is no missing response. HAMD-17 has a total score in a range of 0 (not present) to 52 (severe). Values at Day 0, Week 0 was considered as Baseline value. Remission was defined as HAMD-17 total scores at end of acute treatment phase (Week 8) <=7.
Time Frame: Up to Week 8
Population: PP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Percentage of Participants | 39.7 | 47.2
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.129, GEE model — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.48 to 1.10]

4. Secondary Outcome: Sustained Response Rate Based on HAMD-17 Total Score
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 total score is calculated by summing the individual response scores if there is no missing response. HAMD-17 has a total score in a range of 0 (not present) to 52 (severe). Values at Day 0, Week 0 was considered as Baseline value. Sustained response was defined as response at end of acute treatment phase and an earlier visit and the decrease from Baseline in non-missing HAMD-17 total scores at all visits between these two visits by at least 40%.
Time Frame: Up to Week 8
Population: PP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Percentage of Participants | 51.6 | 56.3
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.354, GEE model — P-value was estimated from a GEE model with Response based on HADM-17 as response variable and treatment, gender as explanatory variables; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.55 to 1.24]

5. Secondary Outcome: Sustained Remission Rate Based on HAMD-17 Total Score
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 total score is calculated by summing the individual response scores if there is no missing response. HAMD-17 has a total score in a range of 0 (not present) to 52 (severe). Values at Day 0, Week 0 was considered as Baseline value. Sustained remission was defined as remission at end of acute treatment phase and an earlier visit and non-missing HAMD-17 total scores at all visits between these two visits <=8.
Time Frame: Up to Week 8
Population: PP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Percentage of Participants | 25.5 | 28.6
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.489, GEE model — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.54 to 1.34]

6. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Weeks 1, 2, 4, 6 and 8
Description: MADRS is a 10-point rating scale. Each item is scored on a scale of 0-6, with a total score range of 0-60. Higher score indicates worst symptoms. This scale is mainly used to assess the efficacy of antidepressant treatment. The ratings were based on the signs and symptoms during the preceding week prior to the visit. Values at Day0, Week 0 was considered as Baseline value. The observed MADRS total score was considered as missing if any item is missing. Change from Baseline in MADRS was obtained by subtracting the Baseline value from the specific post-Baseline value. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -3.6 (0.34) | -3.8 (0.33)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -7.0 (0.47) | -8.3 (0.45)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -11.2 (0.58) | -12.4 (0.56)
  Week 6, n=183, 196: number analyzed (Participants) | 183 | 196
  Week 6, n=183, 196 | -15.5 (0.59) | -16.3 (0.57)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -18.6 (0.57) | -19.5 (0.55)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.627, Mixed model repeated measures analysis — Analysis included Baseline MADRS total score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.70 to 1.16] — Week 1. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.037, Mixed model repeated measures analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.08 to 2.66] — Week 2. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.143, Mixed model repeated measures analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.40 to 2.78] — Week 4. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.330, Mixed model repeated measures analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.81 to 2.40] — Week 6. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.278, Mixed model repeated measures analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.69 to 2.40] — Week 8. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates

7. Secondary Outcome: Change From Baseline in HAMD-17 Depressed Mood Subscale Score (Score of Item 1) at Weeks 1, 2, 4, 6 and 8
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 Depressed Mood Subscale is a factor score of item-1 (Depressed Mood) of HAMD-17 scale. This subscale has a score in a range of 0 (absence of depressed mood feelings) to 4 (when participants report virtually only these feeling states in his/her spontaneous verbal and non-verbal communicationtotal score). Values at Day 0, Week 0 was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline response from the specific post-Baseline response. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -0.4 (0.04) | -0.4 (0.04)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -0.7 (0.06) | -0.8 (0.05)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -1.1 (0.06) | -1.3 (0.06)
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | -1.5 (0.06) | -1.6 (0.06)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -1.9 (0.06) | -1.9 (0.06)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.579, Mixed model repeated measures analysis — Analysis included Baseline HAMD-17 depressed mood subscale score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.09 to 0.16] — Comparison for Week 1. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.163, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.04 to 0.26] — Comparison for Week 2. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.050, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.00 to 0.34] — Comparison for Week 4. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.337, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.09 to 0.26] — Comparison for Week 6. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.714, Mixed model repeated measures analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.14 to 0.20] — Comparison for Week 8. OC dataset was used, where available data at a given time point was used with no missing values filled in with estimates

8. Secondary Outcome: Change From Baseline in HAMD-17 Anxiety/Somatization Subscale Score (Sum of Scores of Items 10, 11, 12, 13, 15 and 17) at Weeks 1, 2, 4, 6 and 8
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 Anxiety/Somatization subscale score was derived as sum of scores of items 10, 11, 12, 13, 15 and 17 from HAMD-17. This subscale has a score in a range of 0 (absence of condition) to 18 (most severe condition). Values at Day 0, Week 0 was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline response from the specific post-Baseline response. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -1.3 (0.12) | -1.1 (0.12)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -2.0 (0.15) | -2.4 (0.14)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -3.0 (0.19) | -3.4 (0.18)
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | -4.0 (0.17) | -4.4 (0.17)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -4.8 (0.16) | -5.1 (0.16)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.358, Mixed model repeated measures analysis — Analysis included Baseline HAMD-17 anxiety/somatization subscale score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.50 to 0.18] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.081, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.04 to 0.75] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.062, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.02 to 0.99] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.118, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.10 to 0.85] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.252, Mixed model repeated measures analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.19 to 0.71] — [estimate comment as in outcome 7, analysis 5]

9. Secondary Outcome: Change From Baseline in HAMD-17 Retardation Subscale Score (Sum of Scores of Items 1, 7, 8 and 14) at Weeks 1, 2, 4, 6 and 8
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 Retardation subscale score was derived as sum of scores of items 1, 7, 8 and 14 from HAMD-17. This subscale has a score in a range of 0 (absence of condition) to 14 (most severe condition). Values at Day 0, Week 0 was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline response from the specific post-Baseline response. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -1.0 (0.10) | -1.0 (0.10)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -1.8 (0.13) | -2.0 (0.13)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -2.9 (0.15) | -3.1 (0.15)
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | -3.9 (0.16) | -3.9 (0.16)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -4.7 (0.17) | -4.9 (0.16)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.573, Mixed model repeated measures analysis — Analysis included Baseline HAMD-17 Retardation subscale score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.20 to 0.35] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.209, Mixed model repeated measures analysis — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.13 to 0.58] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.427, Mixed model repeated measures analysis — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.25 to 0.58] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.851, Mixed model repeated measures analysis — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.40 to 0.48] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.370, Mixed model repeated measures analysis — [p-value comment as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.25 to 0.66] — [estimate comment as in outcome 7, analysis 5]

10. Secondary Outcome: Change From Baseline in HAMD-17 Sleep Disorder Subscale Score (Sum of Scores of Items 4, 5 and 6) at Weeks 1, 2, 4, 6 and 8
Description: HAMD-17 is an extensively used tool to assess the severity of depression and symptom improvement during the treatment. The HAMD-17 adopted for this study consisted of 17 questions with multiple choice responses, each of which is numerically scored. The HAMD-17 Sleep Disorder subscale score was derived as sum of scores of items 4, 5 and 6 from HAMD-17. This subscale has a score in a range of 0 (absence of condition) to 6 (most severe condition). Values at Day 0, Week 0 was considered as Baseline value. Change from Baseline was calculated by subtracting the Baseline response from the specific post-Baseline response. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -0.6 (0.10) | -0.7 (0.09)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -0.8 (0.11) | -1.2 (0.10)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -1.4 (0.11) | -1.6 (0.11)
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | -1.8 (0.11) | -2.0 (0.11)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -2.3 (0.11) | -2.4 (0.11)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.438, Mixed model repeated measures analysis — Analysis included Baseline HAMD-17 Sleep Disorder subscale score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.16 to 0.37] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.014, Mixed model repeated measures analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.07 to 0.66] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.207, Mixed model repeated measures analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.11 to 0.50] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.137, Mixed model repeated measures analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.07 to 0.54] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.299, Mixed model repeated measures analysis — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.14 to 0.46] — [estimate comment as in outcome 7, analysis 5]

11. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness Scale (CGI-S) Score at Weeks 1, 2, 4, 6 and 8
Description: CGI-S records the severity of illness at specific time points, with a range of responses from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Participants with zero values (0) representing "Not assessed" were excluded from analysis. Values at Day 0, Week 0 was considered as Baseline value. Change from Baseline was obtained by subtracting the Baseline value from the specific post-Baseline value. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Scores on a scale
  Week 1, n=184, 199 | -0.3 (0.04) | -0.4 (0.04)
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | -0.7 (0.05) | -0.8 (0.05)
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | -1.1 (0.07) | -1.3 (0.06)
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | -1.6 (0.07) | -1.7 (0.07)
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | -2.1 (0.07) | -2.2 (0.07)
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.804, Mixed model repeated measures analysis — Analysis included Baseline CGI-S score as covariate, treatment, gender, visit and treatment-visit interaction as fixed effects. Unstructured covariance matrix was used; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.10 to 0.13] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.079, Mixed model repeated measures analysis — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.02 to 0.28] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.036, Mixed model repeated measures analysis — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.01 to 0.38] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.248, Mixed model repeated measures analysis — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.08 to 0.31] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.110, Mixed model repeated measures analysis — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.04 to 0.35] — [estimate comment as in outcome 7, analysis 5]

12. Secondary Outcome: Percentage of Participants With a Clinical Global Impression Global Improvement (CGI-I) Score of 1 ("Very Much Improved") or 2 ("Much Improved") at Weeks 1, 2, 4, 6 and 8
Description: For CGI-I rating, the raters indicated their assessment of the participant's total improvement or worsening compared to the participant's condition at the Baseline visit, whether or not the improvement or worsening was thought to be treatment related. Scores ranges from 0 to 7 where 0 represents "Not assessed", and the remaining values 1-7 represent "Very much improved" (1) to "Very much worse" (7). Participants with score 0 were excluded from analysis. All participants in the PP population were analyzed and n=X in the category titles represented the number of participants with data available at the specified time points.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6 and 8
Population: PP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 184 | 199
Percentage of Participants
  Week 1, n=184, 199 | 6 | 7.5
  Week 2, n=182, 199: number analyzed (Participants) | 182 | 199
  Week 2, n=182, 199 | 21.4 | 22.1
  Week 4, n=184, 198: number analyzed (Participants) | 184 | 198
  Week 4, n=184, 198 | 38.6 | 52.5
  Week 6, n=183, 197: number analyzed (Participants) | 183 | 197
  Week 6, n=183, 197 | 67.8 | 71.6
  Week 8, n=176, 188: number analyzed (Participants) | 176 | 188
  Week 8, n=176, 188 | 80.7 | 83.5
Statistical Analysis 1: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.545, GEE model repeated measures — P-value was estimated from a GEE model repeated measures with CGI-I score of 1 or 2 as response variable and treatment, gender as explanatory variables; Odds Ratio, log = 0.78, 95% CI 2-sided [0.35 to 1.75] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.822, GEE model repeated measures — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.58 to 1.54] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.007, GEE model repeated measures — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.38 to 0.86] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.417, GEE model repeated measures — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.54 to 1.29] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: Bupropion XL vs Escitalopram; Test type: Other; p = 0.485, GEE model repeated measures — [p-value comment as in outcome 12, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.49 to 1.40] — [estimate comment as in outcome 7, analysis 5]

13. Secondary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) and Any Serious AE (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Participants who received any of the study treatment and had any non-serious AE or SAE were considered for analysis. Safety Population comprised of all participants who took at least one dose of the study medication.
Time Frame: Up to Week 10
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Participants
  Any non-serious AE | 151 | 150
  Any SAE | 10 | 11

14. Secondary Outcome: Change From Baseline in Hemoglobin, Total Protein, Albumin and Mean Corpuscle Hemoglobin Concentration (MCHC) at the Indicated Time Points
Description: Blood samples were collected at Screening (within 14 days prior to dosing) and at Week 8, Taper visit (Week 9) and Follow-up visit (Week 10). Baseline was considered as the value obtained at Screening. Change from Baseline was calculated by subtracting the Baseline value from the specific post-Baseline values. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per Liter (G/L)
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Gram per Liter (G/L)
  Hemoglobin, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  Hemoglobin, Week 8, n=176, 183 | -0.22 (7.621) | -1.16 (7.874)
  Hemoglobin, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Hemoglobin, Taper, n=13, 16 | -1.54 (5.868) | 1.38 (8.057)
  Hemoglobin, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Hemoglobin, Follow-up, n=10, 8 | -3.10 (12.449) | 0.38 (6.163)
  Total protein, Week 8, n=174, 183: number analyzed (Participants) | 174 | 183
  Total protein, Week 8, n=174, 183 | -0.640 (5.2784) | -0.891 (4.0339)
  Total protein, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  Total protein, Taper, n=12, 15 | 1.197 (6.9347) | 2.000 (8.7513)
  Total protein, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  Total protein, Follow-up, n=8, 12 | -4.650 (5.5131) | -1.227 (4.8619)
  Albumin, Week 8, n=175, 183: number analyzed (Participants) | 175 | 183
  Albumin, Week 8, n=175, 183 | -0.254 (3.0207) | -0.678 (2.8483)
  Albumin, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  Albumin, Taper, n=12, 15 | -0.086 (3.9688) | -0.027 (4.2372)
  Albumin, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  Albumin, Follow-up, n=8, 12 | -1.925 (2.0084) | -1.577 (3.6313)
  MCHC, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  MCHC, Week 8, n=176, 183 | -0.09 (8.933) | 0.76 (9.821)
  MCHC, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  MCHC, Taper, n=13, 16 | 0.54 (8.828) | 2.25 (9.030)
  MCHC, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  MCHC, Follow-up, n=10, 8 | -2.10 (9.398) | -2.88 (5.055)

15. Secondary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Proportion of red blood cells in blood
  Hematocrit, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  Hematocrit, Week 8, n=176, 183 | 0.0016 (0.06088) | -0.0044 (0.02587)
  Hematocrit, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Hematocrit, Taper, n=13, 16 | -0.0051 (0.02105) | 0.0017 (0.02601)
  Hematocrit, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Hematocrit, Follow-up, n=10, 8 | -0.0076 (0.04403) | 0.0051 (0.01509)

16. Secondary Outcome: Change From Baseline in White Blood Cell (WBC) Count, Total Neutrophil, Lymphocyte, Basophil, Eosinophil, Monocyte and Platelet Count at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter (GI/L)
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Giga cells per liter (GI/L)
  WBC count, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  WBC count, Week 8, n=176, 183 | -0.032 (1.6278) | -0.073 (1.6282)
  WBC count, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  WBC count, Taper, n=13, 16 | 0.065 (1.5513) | -0.715 (1.8547)
  WBC count, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  WBC count, Follow-up, n=10, 8 | -0.743 (1.4455) | 0.427 (0.9032)
  Total Neutrophils, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  Total Neutrophils, Week 8, n=176, 183 | 0.101 (1.4835) | -0.165 (1.5540)
  Total Neutrophils, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Total Neutrophils, Taper, n=13, 16 | 0.306 (1.6222) | -0.772 (1.5656)
  Total Neutrophils, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Total Neutrophils, Follow-up, n=10, 8 | -0.869 (1.4578) | 0.424 (0.7470)
  Lymphocytes, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  Lymphocytes, Week 8, n=176, 183 | -0.154 (0.4833) | 0.072 (0.4190)
  Lymphocytes, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Lymphocytes, Taper, n=13, 16 | -0.242 (0.4843) | 0.077 (0.5053)
  Lymphocytes, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Lymphocytes, Follow-up, n=10, 8 | 0.042 (0.3937) | 0.022 (0.4388)
  Basophil, Week 8, n=176, 182: number analyzed (Participants) | 176 | 182
  Basophil, Week 8, n=176, 182 | 0.001 (0.0173) | 0.002 (0.0218)
  Basophil, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Basophil, Taper, n=13, 16 | 0.001 (0.0091) | 0.001 (0.0131)
  Basophil, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Basophil, Follow-up, n=10, 8 | -0.003 (0.0163) | -0.012 (0.0087)
  Eosinophil, Week 8, n=176, 182: number analyzed (Participants) | 176 | 182
  Eosinophil, Week 8, n=176, 182 | -0.004 (0.0788) | 0.010 (0.0899)
  Eosinophil, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Eosinophil, Taper, n=13, 16 | -0.012 (0.0592) | 0.006 (0.0488)
  Eosinophil, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Eosinophil, Follow-up, n=10, 8 | -0.005 (0.0627) | 0.019 (0.0813)
  Monocyte, Week 8, n=176, 182: number analyzed (Participants) | 176 | 182
  Monocyte, Week 8, n=176, 182 | 0.021 (0.1180) | 0.003 (0.1113)
  Monocyte, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Monocyte, Taper, n=13, 16 | -0.001 (0.1023) | -0.031 (0.0917)
  Monocyte, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Monocyte, Follow-up, n=10, 8 | 0.058 (0.1292) | 0.010 (0.0920)
  Platelet count, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  Platelet count, Week 8, n=176, 183 | 7.73 (32.725) | 0.56 (29.492)
  Platelet count, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  Platelet count, Taper, n=13, 16 | 17.15 (35.126) | 7.19 (22.448)
  Platelet count, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  Platelet count, Follow-up, n=10, 8 | 28.50 (35.600) | 5.38 (24.784)

17. Secondary Outcome: Change From Baseline in Total Bilirubin, Direct Bilirubin and Creatinine at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Micromoles per liter (µmol/L)
  Total bilirubin, Week 8, n=175, 181: number analyzed (Participants) | 175 | 181
  Total bilirubin, Week 8, n=175, 181 | -0.812 (4.7591) | -0.071 (4.8022)
  Total bilirubin, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  Total bilirubin, Taper, n=12, 15 | -3.457 (6.5521) | 1.198 (3.9442)
  Total bilirubin, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  Total bilirubin, Follow-up, n=8, 12 | 0.382 (4.0151) | 0.338 (3.4710)
  Direct bilirubin, Week 8, n=175, 180: number analyzed (Participants) | 175 | 180
  Direct bilirubin, Week 8, n=175, 180 | -0.072 (1.3659) | -0.006 (1.2310)
  Direct bilirubin, Taper, n=11, 15: number analyzed (Participants) | 11 | 15
  Direct bilirubin, Taper, n=11, 15 | -1.554 (3.7607) | 0.654 (1.7145)
  Direct bilirubin, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  Direct bilirubin, Follow-up, n=8, 12 | -0.102 (1.1192) | 0.382 (0.9070)
  Creatinine, Week 8, n=174, 183: number analyzed (Participants) | 174 | 183
  Creatinine, Week 8, n=174, 183 | 7.507 (10.6852) | 0.307 (9.0811)
  Creatinine, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  Creatinine, Taper, n=12, 15 | 6.675 (6.9134) | 0.880 (10.3281)
  Creatinine, Follow-up, n=8, 11: number analyzed (Participants) | 8 | 11
  Creatinine, Follow-up, n=8, 11 | 4.237 (8.9291) | 1.618 (9.6668)

18. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transpeptidase (GGT) and Lactose Dehydrogenase (LD) at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
International Units per liter (IU/L)
  ALT, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  ALT, Week 8, n=176, 183 | 2.254 (14.7208) | 1.315 (10.3019)
  ALT, Taper, n=12, 16: number analyzed (Participants) | 12 | 16
  ALT, Taper, n=12, 16 | 7.993 (17.5985) | -1.812 (15.1544)
  ALT, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  ALT, Follow-up, n=8, 12 | -7.337 (21.7809) | 5.938 (19.8234)
  ALP, Week 8, n=176, 181: number analyzed (Participants) | 176 | 181
  ALP, Week 8, n=176, 181 | 1.866 (13.2776) | 0.407 (11.7870)
  ALP, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  ALP, Taper, n=12, 15 | 3.674 (11.5803) | 3.480 (19.2823)
  ALP, Follow-up, n=7, 12: number analyzed (Participants) | 7 | 12
  ALP, Follow-up, n=7, 12 | 5.643 (9.2858) | -3.953 (11.6377)
  AST, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  AST, Week 8, n=176, 183 | 0.330 (7.6259) | 1.099 (6.1029)
  AST, Taper, n=12, 16: number analyzed (Participants) | 12 | 16
  AST, Taper, n=12, 16 | 3.193 (7.4990) | 0.381 (6.0938)
  AST, Follow-up, n=8, 12: number analyzed (Participants) | 8 | 12
  AST, Follow-up, n=8, 12 | 0.925 (23.3485) | 2.867 (11.0264)
  GGT, Week 8, n=175, 181: number analyzed (Participants) | 175 | 181
  GGT, Week 8, n=175, 181 | 0.688 (17.0699) | -0.694 (11.1878)
  GGT, Taper, n=12, 15: number analyzed (Participants) | 12 | 15
  GGT, Taper, n=12, 15 | 1.403 (6.2977) | -3.133 (4.8019)
  GGT, Follow-up, n=7, 12: number analyzed (Participants) | 7 | 12
  GGT, Follow-up, n=7, 12 | -2.029 (5.9637) | 3.916 (25.9888)
  LD, Week 8, n=176, 182: number analyzed (Participants) | 176 | 182
  LD, Week 8, n=176, 182 | 1.292 (32.4627) | 2.879 (27.3838)
  LD, Taper, n=13, 13: number analyzed (Participants) | 13 | 13
  LD, Taper, n=13, 13 | 14.463 (28.9571) | -8.092 (55.0095)
  LD, Follow-up, n=8, 10: number analyzed (Participants) | 8 | 10
  LD, Follow-up, n=8, 10 | 11.037 (45.3316) | -4.150 (33.8871)

19. Secondary Outcome: Change From Baseline in Calcium, Chloride, Cholesterol, Glucose, Potassium, Sodium, Triglyceride and Urea at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Millimole per liter (mmol/L)
  Calcium, Week 8, n=173, 183: number analyzed (Participants) | 173 | 183
  Calcium, Week 8, n=173, 183 | -0.017 (0.1139) | -0.020 (0.1225)
  Calcium, Taper, n=12, 12: number analyzed (Participants) | 12 | 12
  Calcium, Taper, n=12, 12 | -0.019 (0.1906) | 0.012 (0.1091)
  Calcium, Follow-up, n=8, 11: number analyzed (Participants) | 8 | 11
  Calcium, Follow-up, n=8, 11 | -0.060 (0.1032) | -0.060 (0.1352)
  Chloride, Week 8, n=173, 182: number analyzed (Participants) | 173 | 182
  Chloride, Week 8, n=173, 182 | 0.259 (2.7943) | -0.293 (2.5913)
  Chloride, Taper, n=10, 13: number analyzed (Participants) | 10 | 13
  Chloride, Taper, n=10, 13 | -0.498 (3.2001) | -0.566 (2.4684)
  Chloride, Follow-up, n=8, 8: number analyzed (Participants) | 8 | 8
  Chloride, Follow-up, n=8, 8 | -0.287 (3.6588) | -0.178 (4.6453)
  Cholesterol, Week 8, n=175, 181: number analyzed (Participants) | 175 | 181
  Cholesterol, Week 8, n=175, 181 | -0.122 (0.5855) | 0.051 (0.5931)
  Cholesterol, Taper, n=12, 14: number analyzed (Participants) | 12 | 14
  Cholesterol, Taper, n=12, 14 | 0.022 (0.5891) | 0.082 (0.5991)
  Cholesterol, Follow-up, n=9, 11: number analyzed (Participants) | 9 | 11
  Cholesterol, Follow-up, n=9, 11 | -0.124 (0.5149) | -0.122 (0.5899)
  Glucose, Week 8, n=173, 181: number analyzed (Participants) | 173 | 181
  Glucose, Week 8, n=173, 181 | -0.051 (0.6327) | -0.050 (0.5871)
  Glucose, Taper, n=12, 16: number analyzed (Participants) | 12 | 16
  Glucose, Taper, n=12, 16 | 0.352 (0.3822) | 0.106 (0.9661)
  Glucose, Follow-up, n=9, 11: number analyzed (Participants) | 9 | 11
  Glucose, Follow-up, n=9, 11 | -0.194 (0.4089) | 0.025 (1.2117)
  Potassium, Week 8, n=173, 182: number analyzed (Participants) | 173 | 182
  Potassium, Week 8, n=173, 182 | -0.021 (0.3504) | 0.009 (0.3552)
  Potassium, Taper, n=10, 13: number analyzed (Participants) | 10 | 13
  Potassium, Taper, n=10, 13 | -0.114 (0.4165) | 0.046 (0.5095)
  Potassium, Follow-up, n=8, 8: number analyzed (Participants) | 8 | 8
  Potassium, Follow-up, n=8, 8 | -0.110 (0.6221) | 0.036 (0.6556)
  Sodium, Week 8, n=173, 182: number analyzed (Participants) | 173 | 182
  Sodium, Week 8, n=173, 182 | -0.205 (2.4757) | -0.178 (2.5481)
  Sodium, Taper, n=10, 13: number analyzed (Participants) | 10 | 13
  Sodium, Taper, n=10, 13 | -0.611 (3.0799) | 0.978 (1.5853)
  Sodium, Follow-up, n=8, 8: number analyzed (Participants) | 8 | 8
  Sodium, Follow-up, n=8, 8 | -0.175 (3.9085) | 0.770 (3.6011)
  Triglycerides, Week 8, n=175, 181: number analyzed (Participants) | 175 | 181
  Triglycerides, Week 8, n=175, 181 | 0.003 (1.0499) | 0.022 (0.5844)
  Triglycerides, Taper, n=13, 15: number analyzed (Participants) | 13 | 15
  Triglycerides, Taper, n=13, 15 | -0.032 (0.4359) | 0.574 (2.0355)
  Triglycerides, Follow-up, n=9, 11: number analyzed (Participants) | 9 | 11
  Triglycerides, Follow-up, n=9, 11 | 0.637 (1.4045) | 0.181 (0.7767)
  Urea, Week 8, n=174, 183: number analyzed (Participants) | 174 | 183
  Urea, Week 8, n=174, 183 | -0.068 (1.3282) | 0.015 (1.1723)
  Urea, Taper, n=12, 16: number analyzed (Participants) | 12 | 16
  Urea, Taper, n=12, 16 | 0.517 (0.9249) | -0.269 (1.0223)
  Urea, Follow-up, n=8, 11: number analyzed (Participants) | 8 | 11
  Urea, Follow-up, n=8, 11 | 0.687 (0.6998) | -0.419 (1.0801)

20. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Picograms
  MCH, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  MCH, Week 8, n=176, 183 | -0.032 (0.7431) | 0.049 (0.7052)
  MCH, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  MCH, Taper, n=13, 16 | 0.269 (0.7941) | 0.262 (0.7571)
  MCH, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  MCH, Follow-up, n=10, 8 | -0.050 (1.1909) | -0.250 (0.4598)

21. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Femtoliter
  MCV, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  MCV, Week 8, n=176, 183 | 4.668 (62.5158) | -0.090 (2.4759)
  MCV, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  MCV, Taper, n=13, 16 | 0.508 (2.2291) | 0.181 (2.1201)
  MCV, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  MCV, Follow-up, n=10, 8 | 0.320 (3.3565) | 0.287 (1.1205)

22. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at the Indicated Time Points
Description: as for outcome 14
Time Frame: Up to Week 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
10^12 cells per liter
  RBC Count, Week 8, n=176, 183: number analyzed (Participants) | 176 | 183
  RBC Count, Week 8, n=176, 183 | -0.009 (0.2711) | -0.049 (0.2563)
  RBC Count, Taper, n=13, 16: number analyzed (Participants) | 13 | 16
  RBC Count, Taper, n=13, 16 | -0.088 (0.1599) | -0.007 (0.2560)
  RBC Count, Follow-up, n=10, 8: number analyzed (Participants) | 10 | 8
  RBC Count, Follow-up, n=10, 8 | -0.132 (0.4018) | 0.036 (0.1859)

23. Secondary Outcome: Number of Participants With Urinalysis Data Outside the Normal Range
Description: Urine samples were collected at Screening (within 14 days prior to dosing) and at Week 8, Taper visit (Week 9) and Follow-up visit (Week 10). Number of participants with urine specific gravity and potential of hydrogen (pH) outside (higher or lower) the normal range are presented. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 10
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 266 | 268
Participants
  Urine specific gravity, high,Screening, n=265, 255: number analyzed (Participants) | 265 | 255
  Urine specific gravity, high,Screening, n=265, 255 | 20 | 12
  Urine specific gravity, low,Screening, n=265, 255: number analyzed (Participants) | 265 | 255
  Urine specific gravity, low,Screening, n=265, 255 | 1 | 1
  Urine specific gravity,high, Week 8, n=171, 173: number analyzed (Participants) | 171 | 173
  Urine specific gravity,high, Week 8, n=171, 173 | 9 | 7
  Urine specific gravity,low, Week 8, n=171, 173: number analyzed (Participants) | 171 | 173
  Urine specific gravity,low, Week 8, n=171, 173 | 0 | 1
  Urine specific gravity, high, Taper, n=18, 28: number analyzed (Participants) | 18 | 28
  Urine specific gravity, high, Taper, n=18, 28 | 0 | 0
  Urine specific gravity, low, Taper, n=18, 28: number analyzed (Participants) | 18 | 28
  Urine specific gravity, low, Taper, n=18, 28 | 0 | 1
  Urine specific gravity, high, Follow-up, n=7, 14: number analyzed (Participants) | 7 | 14
  Urine specific gravity, high, Follow-up, n=7, 14 | 0 | 3
  Urine specific gravity, low, Follow-up, n=7, 14: number analyzed (Participants) | 7 | 14
  Urine specific gravity, low, Follow-up, n=7, 14 | 0 | 0
  Urine pH, high, Screening, n=265, 266: number analyzed (Participants) | 265 | 266
  Urine pH, high, Screening, n=265, 266 | 7 | 18
  Urine pH, low, Screening, n=265, 266: number analyzed (Participants) | 265 | 266
  Urine pH, low, Screening, n=265, 266 | 37 | 28
  Urine pH, high, Week 8, n=172, 178: number analyzed (Participants) | 172 | 178
  Urine pH, high, Week 8, n=172, 178 | 5 | 9
  Urine pH, low, Week 8, n=172, 178: number analyzed (Participants) | 172 | 178
  Urine pH, low, Week 8, n=172, 178 | 23 | 20
  Urine pH, high, Taper, n=18, 28: number analyzed (Participants) | 18 | 28
  Urine pH, high, Taper, n=18, 28 | 0 | 1
  Urine pH, low, Taper, n=18, 28: number analyzed (Participants) | 18 | 28
  Urine pH, low, Taper, n=18, 28 | 2 | 2
  Urine pH, high, Follow-up, n=7, 14: number analyzed (Participants) | 7 | 14
  Urine pH, high, Follow-up, n=7, 14 | 0 | 0
  Urine pH, low, Follow-up, n=7, 14: number analyzed (Participants) | 7 | 14
  Urine pH, low, Follow-up, n=7, 14 | 2 | 2

24. Secondary Outcome: Number of Participants With Vital Sign Parameters Outside the Clinical Concern Range
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) were taken at Screening (within 14 days prior to dosing), randomization visit (Week 0) and at Weeks 1, 2, 4, 6, 8, Taper visit (Week 9) and Follow-up visit (Week 10). SBP <30 or >170 millimeter of mercury (mmHg); DBP <20 or >110 mmHg and heart rate <40 or >120 beats per minute (bpm) were considered as values outside of clinical concern range and were presented as 'High' or 'Low' values. Number of participants with vital signs outside of clinical concern range at any post-Baseline visit are presented. Only those participants with data available at the specified time points were analyzed.
Time Frame: Up to Week 10
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 260 | 253
Participants
  SBP, high, Any visit post-Baseline | 1 | 0
  SBP, low,Any visit post-Baseline | 0 | 0
  DBP, high, Any visit post-Baseline | 0 | 0
  DBP, low, Any visit post-Baseline | 0 | 0
  HR, high, Any visit post-Baseline | 0 | 1
  HR, low, Any visit post-Baseline | 0 | 0

25. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Outside the Clinical Concern Range
Description: ECG was recorded at Screening (within 14 days prior to dosing) and at Week 8, Taper visit (Week 9) and Follow-up visit (Week 10). PR interval <110 or >220 millisecond (msec); QRS interval <60 or >120 msec and corrected QT (QTc) interval >450 msec were considered as values outside of clinical concern range and were presented as 'High' or 'Low' values. Number of participants with ECG data outside of clinical concern range at any post-Baseline visit are presented. Only those participants with data available at the specified time points were analyzed.
Time Frame: Up to Week 10
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 224 | 222
Participants
  PR interval, high, Any visit post-randomization | 0 | 0
  PR interval, low,Any visit post-randomization | 5 | 2
  QRS interval, high, Any visit post-randomization | 2 | 3
  QRS interval, low, Any visit post-randomization | 0 | 1
  QTc interval, high, Any visit post-randomization | 1 | 3
  QTc interval, low, Any visit post-randomization | 0 | 0

26. Secondary Outcome: Change From Baseline in Changes in Sexual Function Questionnaire (CSFQ)
Description: CSFQ is a questionnaire about sexual activity and sexual function (sexual intercourse, masturbation, sexual fantasies and other activity). CSFQ is a gender-specific questionnaire. Both male and female versions consist of 14 items, each with 5 possible answers. CSFQ has a score in a range of 14 to 70. Higher score indicates higher sexual activity and sexual function. Value at Day 0 (Week 0) was considered as Baseline value. Change from Baseline at Week 8 was calculated by subtracting the Baseline score from the specific post-Baseline score. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline (Day 0) and Week 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 173 | 179
Scores on a scale | 3.0 (6.47) | 0.9 (7.21)

27. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior During Treatment Assessed by Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. It consists of 10 items, each with two possible answers (yes/no). Suicidal ideation was interpreted if "yes" answer at any time during treatment to any one of the five suicidal ideation questions (item 1-5) on the C-SSRS. Suicidal behavior was interpreted if a "yes" answer at any time during treatment to any one of the five suicidal behavior questions (item 6-10) on the C-SSRS. Suicidal ideation or behavior is interpreted if a "yes" answer at any time during treatment to any one of the ten suicidal ideation and behavior questions (item 1-10) on the C-SSRS. Number of participants with at least one on-treatment C-SSRS assessment were analyzed. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline and up to Taper visit (Week 9)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Bupropion XL | Escitalopram
Number analyzed (Participants) | 255 | 249
Participants
  Suicidal Ideation or Behavior | 50 | 43
  Suicidal Ideation | 50 | 43
  Suicidal Behavior | 2 | 1
  Self-Injurious Behavior, no suicidal attempt | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of study treatment and until the end safety follow-up visit (up to Week 10). SAEs were recorded from the time the consent form is signed until the follow-up visit (up to Week 10).
Description: SAEs and non-serious AEs were reported for the Safety Population which comprised of all participants who took at least one dose of the study medication.
Arm/Group | Bupropion XL | Escitalopram
All-Cause Mortality (participants affected / at risk) | 1/266 | 0/268
Serious Adverse Events (participants affected / at risk) | 10/266 | 11/268
Other Adverse Events (participants affected / at risk) | 151/266 | 150/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion XL (N=266) | Escitalopram (N=268)
Depression (Psychiatric disorders) | 2 | 4
Blood pressure increased (Investigations) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1
Lacrimal structure injury (Injury, poisoning and procedural complications) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion XL (N=266) | Escitalopram (N=268)
Nausea (Gastrointestinal disorders) | 28 | 50
Dry mouth (Gastrointestinal disorders) | 16 | 15
Constipation (Gastrointestinal disorders) | 14 | 9
Abdominal discomfort (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1
Gastric dilatation (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 25 | 23
Headache (Nervous system disorders) | 20 | 15
Somnolence (Nervous system disorders) | 1 | 13
Tremor (Nervous system disorders) | 8 | 2
Dysgeusia (Nervous system disorders) | 4 | 2
Head discomfort (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 1
Poor quality sleep (Nervous system disorders) | 2 | 1
Anticholinergic syndrome (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Head titubation (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 15 | 13
Urinary tract infection (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Peritonsillitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 2 | 5
Fatigue (General disorders) | 2 | 5
Thirst (General disorders) | 3 | 4
Chest discomfort (General disorders) | 3 | 2
Pyrexia (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 2
Crying (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Hunger (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sensation of foreign body (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 2
Anxiety (Psychiatric disorders) | 5 | 1
Agitation (Psychiatric disorders) | 4 | 1
Dysphoria (Psychiatric disorders) | 2 | 2
Initial insomnia (Psychiatric disorders) | 2 | 2
Hallucination, auditory (Psychiatric disorders) | 1 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Fear (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1
Middle insomnia (Psychiatric disorders) | 1 | 0
Psychiatric symptom (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Blood glucose increased (Investigations) | 1 | 5
White blood cell count decreased (Investigations) | 4 | 1
Heart rate increased (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood pressure increased (Investigations) | 2 | 0
Blood triglycerides increased (Investigations) | 1 | 1
Electrocardiogram T wave abnormal (Investigations) | 2 | 0
Weight increased (Investigations) | 0 | 2
Bilirubin conjugated increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram ST-T change (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Electrocardiogram high voltage (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Lipids abnormal (Investigations) | 1 | 0
Lipoprotein (a) increased (Investigations) | 1 | 0
Lymphocyte percentage increased (Investigations) | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 15
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Palpitations (Cardiac disorders) | 11 | 5
Tachycardia (Cardiac disorders) | 3 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1
Defect conduction intraventricular (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 4 | 2
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 1
Eye pain (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Photopsia (Eye disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
White blood cell disorder (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.